CLINICAL TRIAL: NCT06970613
Title: Effects Of Two Different Methods In Reducing Dental Anxiety In Children: An Experimental Study
Brief Title: Effects Of Two Different Methods In Reducing Dental Anxiety In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melis AKYILDIZ (Other)
Responsible Party: Sponsor-Investigator, Melis AKYILDIZ, Asistant Professor, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADU-DHF-BNSAydogan-01
Record Dates: First submitted 2025-04-20; First posted 2025-05-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Dental Anxiety
Keywords: Pediatric Dental Anxiety; Dental anxiety; Pet Therapy

STUDY DESIGN:
Intervention Model Description: The study is an experimental, controlled randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Watching cartoons (Experimental): Non-pharmacological behavioral guidance techniques and cartoons will be watched as a distraction method.
  Interventions: Behavioral: Watching cartoons
- Robot Cat (Experimental): Non-pharmacological behavioral guidance techniques and a robot cat will be used as a distraction method.
  Interventions: Behavioral: Robot cat

INTERVENTIONS:
Behavioral: Watching cartoons — While watching the cartoons, local anesthesia will be applied and restorative treatments will be completed.
  Arms: Watching cartoons
Behavioral: Robot cat — Local anesthesia will be applied with the robot cat in their lap during the treatment and their restorative treatments will be completed.
  Arms: Robot Cat

SUMMARY:
This study aimed to determine the effects of two different methods in reducing dental anxiety in children. The secondary aim of our research was to determine the levels of dental anxiety in children and the factors that may be related to it.

DETAILED DESCRIPTION:
Anxiety is defined as an emotional state that comes before encountering a feared situation or object. Anxiety can also be seen as a coping mechanism that a person develops to cope with stress, existing before the feared situation actually occurs. Many factors such as physical, cognitive, psychosocial, and economic factors can play a role in the development of anxiety, as well as treatments and interventions related to oral and dental health can be a source of anxiety for the individual. Negative and strong feelings related to any type of dental procedure are called dental anxiety. According to studies, the prevalence of dental anxiety is estimated to vary between 3% and 43% worldwide. Dental anxiety/fear is a very common problem worldwide, observed frequently in children as well as in the elderly, adults, and adolescents.

The prevalence of dental anxiety in children is estimated to be between 5% and 20%. Dental anxiety in children may be due to internal factors such as age and temperament, as well as external factors related to the family such as anxiety and socio-economic status, and external dental factors such as dental-related conditions and medical experiences. In addition, the first dental visit, painful and disturbing stimuli that the child may encounter (such as the instruments used, the waiting room, the doctor's appearance, sounds), the doctor's approach, and the culture in which the child was born and raised are also important factors for dental anxiety.

In order to increase the success of dental treatment in children, determining the level of dental anxiety is important for the application of appropriate techniques. In order to manage dental anxiety in a healthy way and increase the child's compliance with treatment, determining dental anxiety, applying management approaches according to the type and level of dental anxiety, informing children appropriate to their age before any medical interventions and procedures to be performed regarding oral and dental health and using appropriate methods will contribute to controlling the child's worries and fears. In this way, dental anxiety is reduced; It can be effective in reducing the patient's avoidance of dental visits and entering a vicious cycle of dental anxiety, tooth decay/loss, poor oral hygiene, oral and dental health problems that may occur in adulthood and related eating difficulties, pain, avoidance of socialization behaviors and increasing children's compliance with treatment, as well as allowing dentists to work with less stress and minimizing possible time losses. For this reason, recognizing and resolving dental anxiety while still in childhood is an extremely important issue for the success of treatment.

When studies conducted to reduce dental anxiety in children were examined; it was found that distraction through videotapes reduced dental anxiety and fear, and at the same time, it would make working with this patient group, which is more difficult for dentists, more comfortable and would reduce the time spent, while in a study using humanoid robots, a newer technology, it was concluded that robots also helped children cope with dental anxiety and stress, and in another study conducted in a similar way to reduce dental fear in children; it was concluded that informing children by playing with play dough from the dentist's set before the procedure to be performed in dental applications reduced dental anxiety, and that the dental anxiety of the children in the control group who did not play with play dough was higher than before the procedure. Another study has shown that distracting children's attention by playing with toys in the waiting room before a dental procedure can also be effective in reducing dental anxiety.

In a study conducted with adults, it was stated that dog-assisted therapy and dental anxiety were related, that there was a decrease in perceived discomfort during the intervention and that there was an improvement in the patient's evaluation of the experience. Similarly, it has been shown that animal-assisted treatments have positive effects on dental anxiety in children. For this purpose, professional dogs that have received therapy support training are used. However, it has been emphasized that animal-assisted dental treatments can be risky for both the dog and the dental staff due to clinical hygiene conditions and can be applied if the necessary precautions are taken. Today, social robots have been developed thanks to advanced technologies and studies have shown that they are beneficial for individuals who feel the need for emotional support. In this study, it was aimed to investigate the effect of robot cats, which are both suitable for use in hygienic conditions and developed for those who need emotional support, on dental anxiety in children.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 6-10
* Systemically and mentally healthy
* Not allergic to local anesthetics
* Not afraid of pets
* In need of restorative treatment
* No spontaneous pain complaints
* Parents who agreed to participate in the study

Exclusion Criteria:

* Children with previous complaints of severe spontaneous pain
* Teeth requiring endodontic treatment
* Children who are definitely negative according to the Frankl behavior scale

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Modified Child Dental Anxiety Scale (MCDASf) | Baseline (T1)
  It consists of eight questions, each addressing a specific dental procedure or situation. For each question, children are asked to rate their anxiety using a set of five facial expressions, ranging from relaxed/happy to very worried/scared.
  Each face corresponds to a numerical score from 1 to 5:1=Not worried at all,2=A little worried,3=Quite worried,4=Very worried,5=Really worried Children select the face that best matches their feelings for each question. The total score is calculated by summing the scores for all eight items, giving a possible range from 8 to 40:A total score of 8 indicates no dental anxiety. A total score of 40 indicates extreme dental anxiety.
Modified Child Dental Anxiety Scale (MCDASf) | Immediately after the local anaesthesiat (T3)
  It consists of eight questions, each addressing a specific dental procedure or situation. For each question, children are asked to rate their anxiety using a set of five facial expressions, ranging from relaxed/happy to very worried/scared.
  Each face corresponds to a numerical score from 1 to 5:1=Not worried at all,2=A little worried,3=Quite worried,4=Very worried,5=Really worried Children select the face that best matches their feelings for each question. The total score is calculated by summing the scores for all eight items, giving a possible range from 8 to 40:A total score of 8 indicates no dental anxiety. A total score of 40 indicates extreme dental anxiety.

SECONDARY OUTCOMES:
Face, legs, activity, cry, consobility (FLACC) test | During the local anaesthesia (T2)
  Face, legs, activity, cry, consobility (FLACC) test is a behavior rating scale. The Turkish language validity of the pain assessment scale developed by Merkel and colleagues in 1997 and used in the hospital assessment of acute process-related and postoperative pain was done by Şenayli et al. (2006). The measurement is made by evaluating five behavioral categories (facial expression, leg movements, activity, crying, comfortability) in children. Each item is scored between 0 and 2. A score of 0 indicates that the patient is comfortable; 1-3 indicates mild pain; 4-6 indicates moderate pain, and 7-10 indicates severe pain.
Venham Picture Test | Baseline (T1)
  The Venham Picture Test is one of the visual self-report methods used to assess children's anxiety levels, particularly in clinical settings such as dentistry. It consists of eight cards, each displaying two cartoon figures side by side-one depicting a non-worried (relaxed or happy) child and the other depicting a worried (anxious or distressed) child. Each card is numbered and presented in a fixed order.
  Children are asked to look at each pair and select the figure that best represents how they feel at that moment. For each card, if the child chooses the worried figure, they receive a score of 1; if they choose the non-worried figure, they receive a score of 0.The lowest possible total score is 0, indicating no anxiety, where the child consistently chooses the non-worried figures.The highest possible total score is 8, indicating high anxiety, where the child selects the worried figure on all eight cards.
Venham Picture Test | Immediately after the local anaesthesiat (T3)
  The Venham Picture Test is one of the visual self-report methods used to assess children's anxiety levels, particularly in clinical settings such as dentistry. It consists of eight cards, each displaying two cartoon figures side by side-one depicting a non-worried (relaxed or happy) child and the other depicting a worried (anxious or distressed) child. Each card is numbered and presented in a fixed order.
  Children are asked to look at each pair and select the figure that best represents how they feel at that moment. For each card, if the child chooses the worried figure, they receive a score of 1; if they choose the non-worried figure, they receive a score of 0.The lowest possible total score is 0, indicating no anxiety, where the child consistently chooses the non-worried figures.The highest possible total score is 8, indicating high anxiety, where the child selects the worried figure on all eight cards.
Wong-Baker Faces pain rating scale | Immediately after the local anaesthesiat (T3)
  This scale is a pain measurement scale developed for the elderly, children and patient populations with whom communication is difficult, including facial images expressing various emotions. It is frequently preferred, especially for children under the age of six and in the preschool period, due to its repeatability and ease of use. The Wong-Baker Face Scale consists of six cartoon faces, ranked from very happy to very unhappy. Children are asked which shape they find closest to their own feelings and are asked to mark it. The total score according to the scale is calculated by giving 0 to the happiest face and 5 to the unhappiest face.

CONTACTS AND LOCATIONS:
Overall Officials: Rahsan Cevik Akyil, Prof. Dr., Study Director — Aydin Adnan Menderes University; Bahar Melis AKYILDIZ, Phd, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No